CLINICAL TRIAL: NCT00997737
Title: Diaphragm Mobility During Respiratory Exercises With Incentive Spirometry in Healthy Individuals
Brief Title: Diaphragm Activity During Incentive Spirometry and Diaphragmatic Breathing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Wellington Yamaguti, Hospital Sírio Libanês
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSL2008/26
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2009-10

CONDITIONS: Diaphragm Mobility; Breathing Exercises; Incentive Spirometry; Diaphragmatic Breathing
Keywords: incentive spirometry; diaphragm mobility; ultrasound; diaphragmatic breathing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DB, VI and FV (Experimental): Breathing exercises
  Interventions: Device: DB, VI and FI

INTERVENTIONS:
Device: DB, VI and FI — Two modalities of respiratory exercises based on deep and slow inspirations will be used: DB and IS. During DB, the researcher will place one hand slightly below the lower ribs in the abdominal region of the subject and the subject will be instructed to perform inspirations up to the maximum level of volume avoiding rib cage displacement; this recommendation will also be valid for exercises using incentive spirometers. IS will be executed using two different devices: Triflo II and Voldyne.
  Other Names: diaphragmatic exercice; incentive spirometry

SUMMARY:
The objective of the present study is to evaluate diaphragm activity during three breathing exercises: diaphragmatic breathing (DB), flow-oriented (Triflo II)incentive spirometry and volume-oriented (Voldyne) incentive spirometry.

Seventeen healthy subjects will be studied (8 man and 9 woman).

DETAILED DESCRIPTION:
Right diaphragmatic mobility will be evaluated by determining the craniocaudal displacement of the left branch of the portal vein using a B-mode ultrasound device (Logic 500, Pro Series®; General ElectricMedical Systems, Milwaukee, WI, USA). The ultrasound technician will use a 3.5 MHz convex transducer positioned in the right subcostal region, with the incidence angle perpendicular to the craniocaudal axis, in the direction of the inferior vena cava. Next, an intraparenchymal portal branch will be identified in the field of vision and its position will be traced with the curser during the forced inspiration and expiration. The craniocaudal displacement of these points will be considered to be the amount of right diaphragmatic mobility.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 to 40 years old
* Having a normal body mass index
* Being a non-smoker
* Not knowing the DB and the IS techniques
* Reporting the absence of respiratory diseases.

Exclusion Criteria:

* Presenting alteration in respiratory function detected by functional analysis of lung volume and capacity
* Inability to understand or perform the procedure.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
ultrasound evaluation of the diaphragm mobility | six - eight months

SECONDARY OUTCOMES:
pulmonary function test | six - eight months

CONTACTS AND LOCATIONS:
Overall Officials: Wellington P Yamaguti, Master, Principal Investigator — Hospital Sírio-Libanês
Locations (1):
- Instituto de Ensino e Pesquisa do Hospital Sírio Libanês, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Yamaguti WP, Sakamoto ET, Panazzolo D, Peixoto Cda C, Cerri GG, Albuquerque AL. Diaphragmatic mobility in healthy subjects during incentive spirometry with a flow-oriented device and with a volume-oriented device. J Bras Pneumol. 2010 Nov-Dec;36(6):738-45. doi: 10.1590/s1806-37132010000600011. English, Portuguese. PMID 21225177